CLINICAL TRIAL: NCT00981708
Title: A Phase I/II Trial of Lenalidomide Combined With Cyclophosphamide and Intermediate Dose Dexamethasone in Patients With Primary (AL) Systemic Amyloidosis
Brief Title: Lenalidomide, Dexamethasone and Cyclophosphamide in Amyloidosis (AL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Principal Investigator, Meletios A. Dimopoulos, Professor of Medicine, University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-178
Record Dates: First submitted 2009-09-19; First posted 2009-09-22 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; lenalidomide; newly diagnosed; relapsed; primary systemic AL amyloidosis
MeSH Terms: conditions — Amyloidosis; Recurrence; Immunoglobulin Light-chain Amyloidosis | interventions — Lenalidomide; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Lenalidomide, Dexamethasone and cyclophosphamide
  Interventions: Drug: Lenalidomide, Dexamethasone and Cyclophosphamide

INTERVENTIONS:
Drug: Lenalidomide, Dexamethasone and Cyclophosphamide — Lenalidomide capsules on days 1 to 21. the dose starts at 5 mg/day up to 25 mg/day.
  Dexamethasone tablets on days 1 to 4. Dose 20 mg per day.
  Cyclophosphamide tablets on days 1 to 10. The dose starts at 50 mg per day up to 100 mg per day.
  The cycle is to be repeated every 28 days (4 weeks)
  Other Names: Revlimid; Endoxan; Dexamethasone

SUMMARY:
The purpose of this study is to determine the safety and activity of the combination of lenalidomide with intermediate dose dexamethasone and cyclophosphamide in patients with primary systemic (AL ) amyloidosis.

DETAILED DESCRIPTION:
Primary systemic amyloidosis (AL) is a plasma cell dyscrasia where amyloid fibrils are formed by monoclonal immunoglobulin light chains and deposit in various organs causing tissue damage and dysfunction. It is a rare disease with an incidence of 8 patients per million per year. Virtually all patients die of this disease with a median survival of 12-18 months and less than approximately 5% surviving 10 years. The current therapeutic approach to systemic amyloidosis is based on the observation that amyloid deposits can be reabsorbed and organ function can be restored if the concentration of the amyloidogenic precursor is reduced. The recognized standard treatment for patients with amyloidosis is alkylating agent-based chemotherapy - some selected patients can be treated with high dose melphalan with autologous stem cell transplantation. Recent studies have led to an improved understanding of the biology of plasma cells. Interactions between the bone marrow microenvironment and plasma cells have a critical growth regulating influence on myeloma cells. Thalidomide has shown significant activity in multiple myeloma patients with relapsing or refractory disease and even more in newly diagnosed patients. However, thalidomide causes somnolence, fatigue, constipation, and peripheral neuropathy and is not well tolerated in patients with AL amyloidosis. Lenalidomide is a small molecule structurally related to thalidomide with potent immunomodulatory effects. Lenalidomide has been found to be significantly active in relapsed multiple myeloma both in vitro and in Phase I, II and III clinical trials, including patients who had previously failed thalidomide. Unlike thalidomide, lenalidomide causes no significant sedation, constipation, neuropathy, or rash. Deep vein thrombosis ,especially in combination with dexamethasone, has been reported . Combination of thalidomide with with alkylating agents (such as melphalan or cyclophosphamide) have been very active in patients with myeloma and have superior activity than combinations of alkylating agents with steroids alone. However, the toxicity profile of thalidomide is problematic for this combination in patients with AL. combinations of lenalidomide with alkylating agents (Melphalan + prednisone +Lenalidomide)are feasible and very active in patients with multiple myeloma. Cyclophosphamide has a more favorable toxicity profile than melphalan when used in oral combinations with dexamethasone and thalidomide. However, given the remarkable antimyeloma activity of lenalidomide, overall improved toxicity profile of lenalidomide compared with thalidomide and a need for improved treatments for this incurable malignancy, the combinations of lenalidomide are worthy of study. Preliminary data from Mayo clinic using CC-5013 and dexamethasone demonstrates that lenalidomide is tolerable and has activity in patients with AL amyloidosis and may be useful in patients with AL amyloidosis who either are not candidates for high dose chemotherapy and peripheral blood stem cell transplantation or who have failed prior therapies. Efficacy and tolerability of oral cyclophosphamide , combined with dexamethasone and thalidomide, is well documented in patients with refractory or relapsed multiple myeloma while this combination has been used in patients with AL amyloidosis . Intermediate dose dexamethasone is tolerable and without significant toxicity in patients with AL amyloidosis . The combination of alkylating agents with thalidomide and dexamethasone has been effective in patients with AL amyloidosis . The combination of an alkylating agent with Lenalidomide and intermediate dose dexamethasone may lead to more rapid hematologic responses than either agent alone , and subsequently may lead to increased organ response rates . Therefore, in this phase I/II trial we explore the safety and efficacy of the combination of the alkylating agent cyclophosphamide to lenalidomide and intermediate dose dexamethasone in patients who are no candidates for high dose melphalan chemotherapy with autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >=18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Confirmed diagnosis of AL amyloidosis (see appendix 3)
5. Need for treatment in the judgment of their treating physician
6. Evaluable or measurable disease defined by any of the following:

   * Measurable serum free light chains >= 10 mg/dL, kappa or lambda, provided kappa/lambda ratio is abnormal (measurable disease)
   * Monoclonal protein in the serum >= 1 g/dL
7. ECOG Performance Status (PS) 0, 1, 2 or 3
8. Laboratory test results within these ranges:

   * Absolute neutrophil count >= 1.5 x 109/L
   * Platelet count >= 100 x 109/L
   * Serum creatinine >= 2.5 mg/dL
   * Total bilirubin >= 1.5 mg/dL
   * AST (SGOT) and ALT (SGPT) > 2 x ULN or > 5 x ULN if hepatic metastases are present.
9. Women of childbearing potential (WCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10 - 14 days prior to therapy and repeated within 24 hours of starting study drug and must begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. Women must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. (See Appendix 1 Pregnancy Testing Guidelines and Acceptable Birth Control Methods.)
10. Disease free of prior malignancies for >= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
11. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. (patients intolerant to ASA may use low molecular weight heparin).

Exclusion Criteria:

1. Patients with symptomatic multiple myeloma with asymptomatic biopsy confirmed AL amyloidosis (Appendix 3)
2. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
3. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
4. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
5. Use of any other experimental drug or therapy within 28 days of baseline.
6. Known hypersensitivity to thalidomide.
7. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
8. Any prior use of lenalidomide.
9. Concurrent use of other anti-cancer agents or treatments.
10. Known positive for HIV or infectious hepatitis, type A, B or C.
11. > grade 2 peripheral neuropathy
12. Life expectancy < 3 months
13. Concurrent use of steroids (Patients may receive prednisone up to 20 mg/d, or equivalent corticosteroids for concurrent illness or adrenal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-02; Primary Completion 2011-01-11 (Actual); Study Completion 2016-01-11 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated dose of lenalidomide and cyclophosphamide and assess the hematologic response rate of the combination of Cyclophosphamide/Dexamethasone plus lenalidomide in patients with AL amyloidosis. | At month 2 for assesment of maximum tolerated dose and monthly for hematologic response
  Maximum Tolerated Dose

SECONDARY OUTCOMES:
To assess the toxicity of Cyclophosphamide/Dexamethasone plus lenalidomide combination in patients with AL amyloidosis and organ response rate | Monthly for toxicity and every 3-6 months for organ response
  Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Meletios A Dimopoulos, MD, Principal Investigator — University of Athens, School of Medicine
Locations (1):
- Alexandra Hospital , Department of Clinical Therapeutics, Athens, Attica, Greece

REFERENCES:
- [Derived] Gavriatopoulou M, Garcia-Sanz R, Kastritis E, Morel P, Kyrtsonis MC, Michalis E, Kartasis Z, Leleu X, Palladini G, Tedeschi A, Gika D, Merlini G, Sonneveld P, Dimopoulos MA. BDR in newly diagnosed patients with WM: final analysis of a phase 2 study after a minimum follow-up of 6 years. Blood. 2017 Jan 26;129(4):456-459. doi: 10.1182/blood-2016-09-742411. Epub 2016 Nov 21. PMID 27872060
- [Derived] Dimopoulos MA, Garcia-Sanz R, Gavriatopoulou M, Morel P, Kyrtsonis MC, Michalis E, Kartasis Z, Leleu X, Palladini G, Tedeschi A, Gika D, Merlini G, Kastritis E, Sonneveld P. Primary therapy of Waldenstrom macroglobulinemia (WM) with weekly bortezomib, low-dose dexamethasone, and rituximab (BDR): long-term results of a phase 2 study of the European Myeloma Network (EMN). Blood. 2013 Nov 7;122(19):3276-82. doi: 10.1182/blood-2013-05-503862. Epub 2013 Sep 4. PMID 24004667
- [Derived] Kastritis E, Terpos E, Roussou M, Gavriatopoulou M, Pamboukas C, Boletis I, Marinaki S, Apostolou T, Nikitas N, Gkortzolidis G, Michalis E, Delimpasi S, Dimopoulos MA. A phase 1/2 study of lenalidomide with low-dose oral cyclophosphamide and low-dose dexamethasone (RdC) in AL amyloidosis. Blood. 2012 Jun 7;119(23):5384-90. doi: 10.1182/blood-2011-12-396903. Epub 2012 Apr 18. PMID 22517904